CLINICAL TRIAL: NCT00990106
Title: A Placebo-Controlled Augmentation Trial of Prazosin for PTSD
Brief Title: Augmentation Trial of Prazosin for Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT074250; 1P20AA017839-01 (NIH)
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Stress Disorders, Post-Traumatic; Combat Disorders; Sleep Disorders
Keywords: posttraumatic stress disorder; PTSD; nightmares; prazosin; sleep disturbance; combat trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Sleep Wake Disorders; Parasomnias | interventions — Prazosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prazosin hydrochloride (Active Comparator): prazosin Pfizer Minipress
  oral capsules
  Subject will be titrated up to the optimum tolerated dose based on the Dosing Algorithm. Males and females will be titrated differently with females titrated slower and to a lower maximum daily dose.
  Interventions: Drug: prazosin hydrochloride
- placebo (Placebo Comparator): placebo
  oral capsules
  Subject will be titrated up to the optimum tolerated dose based on the Dosing Algorithm. Males and females will be titrated differently with females titrated slower and to a lower maximum daily dose.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prazosin hydrochloride — Subject will be titrated up to the optimum tolerated dose based on the Dosing Algorithm. Males and females will be titrated differently with females titrated slower and to a lower maximum daily dose. The first dose will be taken while the participant is in bed for the night to avoid orthostatic syncope, an uncommon but recognized "first dose" effect of prazosin or any alpha-1 antagonist if started at a high dose. The first dose effect is avoidable by starting treatment with a low dose (1 mg at bedtime) then titrating the dose upward gradually.
  Other Names: prazosin; Pfizer Minipress
  Arms: prazosin hydrochloride
Drug: placebo — placebo
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether prazosin will:

* reduce the incidence of nightmares and sleep disturbance
* increase functioning and sense of well being in combat-trauma exposed Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) Veterans.

DETAILED DESCRIPTION:
This is a 15-week randomized parallel design, double-blind, placebo-controlled augmentation trial of prazosin to evaluate the efficacy and tolerability of prazosin augmentation in the treatment of PTSD trauma-related nightmares, sleep disturbance, global function and sense of well-being, and other clinical features and comorbidities of PTSD. Participants will be 210 OIF/OEF soldiers and veterans who have suffered war zone trauma. Participants will be randomized 1:1 to prazosin or placebo and all previous psychotropic medications and/or psychotherapy will be maintained constant. Randomization will be stratified by site and use of an antidepressant.

ELIGIBILITY:
Inclusion Criteria

* Age >18 years;
* Clear evidence of exposure to one or more war zone trauma events sufficient to satisfy DSM-IV criterion A1 for diagnosis of PTSD;
* DSM-IV diagnosis of PTSD derived from the CAPS; CAPS total score >50;
* CAPS Recurrent Distressing Dreams item score >5 (of maximum score of 8);
* stable dose of non-exclusionary medications and psychotherapeutic treatment for at least 4 weeks prior to randomization;
* good general medical health.
* Female participants must agree to use a reliable form of birth control during the study.

Exclusion Criteria

* Psychiatric/Behavioral - meets DSM-IV criteria for current schizophrenia, schizoaffective disorder, psychotic disorder, delirium, or any DSM-IV cognitive disorder; substance dependence disorder within 3 months or any current substance dependence; current cocaine or stimulant abuse; severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to patient or others.
* Medical - acute or unstable chronic medical illness, including unstable angina, recent myocardial infarction (within 6 months), congestive heart failure, preexisting hypotension or orthostatic hypotension, chronic renal or hepatic failure, pancreatitis, Meniere's disease, benign positional vertigo; narcolepsy, or diagnosed sleep apnea; allergy or previous adverse reaction to prazosin or other alpha-1 antagonist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray Raskind, MD, Study Chair — Department of Veterans Affairs Puget Sound Health Care System
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Raskind MA, Peterson K, Williams T, Hoff DJ, Hart K, Holmes H, Homas D, Hill J, Daniels C, Calohan J, Millard SP, Rohde K, O'Connell J, Pritzl D, Feiszli K, Petrie EC, Gross C, Mayer CL, Freed MC, Engel C, Peskind ER. A trial of prazosin for combat trauma PTSD with nightmares in active-duty soldiers returned from Iraq and Afghanistan. Am J Psychiatry. 2013 Sep;170(9):1003-10. doi: 10.1176/appi.ajp.2013.12081133. PMID 23846759
- [Derived] Raskind MA, Millard SP, Petrie EC, Peterson K, Williams T, Hoff DJ, Hart K, Holmes H, Hill J, Daniels C, Hendrickson R, Peskind ER. Higher Pretreatment Blood Pressure Is Associated With Greater Posttraumatic Stress Disorder Symptom Reduction in Soldiers Treated With Prazosin. Biol Psychiatry. 2016 Nov 15;80(10):736-742. doi: 10.1016/j.biopsych.2016.03.2108. Epub 2016 Apr 11. PMID 27320368

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo: placebo titrated in the same manner as prazosin arm.
Period: Overall Study
Arm/Group | Prazosin Hydrochloride | Placebo
Started | 32 | 35
Completed | 23 | 23
Not Completed | 9 | 12
Not completed — "too busy" to continue | 1 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — opted for open label prazosin | 1 | 1
Not completed — relocation/deployment | 4 | 1
Not completed — started exclusionary medication | 0 | 1
Not completed — planned major surgery | 0 | 1
Not completed — scheduling conflicts | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin Hydrochloride | Placebo | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (6.6) | 30.8 (6.5) | 30.4 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 26 | 31 | 57
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale for DSM-IV (CAPS) Recurrent Distressing Dreams Item
Description: Item B-2 "recurrent distressing dreams of the event" is a single item from the Clinician Administered PTSD Scale. The rating consists of two parts: Frequency and Intensity. Symptom frequency rated 0 to 4. Symptom intensity rated 0 to 4. Frequency plus Intensity ratings equal the total score. A higher score is worse; a lower score is better. This outcome measure evaluates the change in score from Baseline to Week 15.
Time Frame: Baseline to Week 15
Population: Of the 67 subjects randomized, 46 completed the full 15 weeks (23 per group). The outcome data reports only those 46 participants who completed the full 15 weeks.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Prazosin Hydrochloride | Placebo
Number analyzed (Participants) | 23 | 23
Scores on a Scale | 3.1 (0.3) | 1.2 (0.3)

2. Primary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI)
Description: Pittsburgh Sleep Quality Index is a self-report questionnaire assessing sleep quality and disturbances over a 1-month time interval. A global score is obtained by summing the seven component subscales (total score range: 0-21). A score of 5 or less indicates good sleep quality. A score of more than 5 indicates poor sleep quality. Change is measured from Baseline to Week 15.
Time Frame: Baseline to Week 15
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Prazosin Hydrochloride | Placebo
Number analyzed (Participants) | 23 | 23
Scores on a Scale | 5.6 (0.7) [12.8 to 15.5] | 2.8 (0.6) [7.1 to 9.9]

3. Primary Outcome: Clinical Global Impression of Change (CGIC)
Description: The Clinical Global Impression of Change is a 7-point scale that rates global change compared to baseline (1=markedly improved, 2=moderately improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=moderately worse, 7=markedly worse). The CGIC is used to determine the impact of treat effects on meaningful and distinct change in overall sense of well-being and functioning. This outcome measures the proportion of responders who were rated markedly or moderately improved at Week 15 compared to Baseline.
Time Frame: Change from Baseline to Week 15
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Prazosin Hydrochloride | Placebo
Number analyzed (Participants) | 23 | 23
Percentage of responders | 64 [44 to 79] | 27 [14 to 45]

ADVERSE EVENTS:
Arm/Group | Prazosin Hydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 2/35
Other Adverse Events (participants affected / at risk) | 18/32 | 25/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin Hydrochloride (N=32) | Placebo (N=35)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) — One participant hospitalized for suicidal ideation.
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) — One participant took a nonlethal overdose of oxycodone/acetaminophen as a suicide attempt.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin Hydrochloride (N=32) | Placebo (N=35)
syncope (General disorders) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
lack of energy (General disorders) | 0 (0) | 1 (1)
palpitations (Cardiac disorders) | 3 (3) | 1 (1)
drowsiness (General disorders) | 1 (1) | 3 (3)
depression (Psychiatric disorders) | 0 (0) | 2 (2)
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
headache (General disorders) | 1 (1) | 8 (8)
dizziness (General disorders) | 9 (10) | 7 (7)
nausea (Gastrointestinal disorders) | 5 (5) | 6 (7)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
other (General disorders) | 18 (35) | 25 (42)

LIMITATIONS AND CAVEATS:
The sample was restricted to soldiers with frequent recalled combat trauma nightmares. More studies in civilian trauma PTSD are needed. Results cannot be extrapolated to persons with PTSD who do not recall trauma nightmares.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No